CLINICAL TRIAL: NCT00417482
Title: Antipsychotic Discontinuation in Alzheimer's Disease
Acronym: ADAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #5598R; 5R01AG021488 (NIH)
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-03

CONDITIONS: Alzheimer Disease; Psychotic Disorders; Agitation; Aggression
Keywords: Risperidone treatment, psychosis, agitation, aggression,; discontinuation, placebo
MeSH Terms: conditions — Alzheimer Disease; Psychotic Disorders; Psychomotor Agitation; Aggression | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Risperidone-risperidone (Other): Risperidone for 16 weeks followed by risperidone for 16 weeks
  Interventions: Drug: risperidone
- Risperidone-Placebo (Other): Risperidone for 16 weeks followed by placebo for 16 weeks
  Interventions: Drug: risperidone
- Placebo-Placebo (Other): Placebo for 16 weeks followed by placebo for 16 weeks
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — Risperidone open label flexible dose 0.25 to 3 mg daily for first 16 weeks; dose at 16 weeks then fixed for randomized trial
  Other Names: Risperdal

SUMMARY:
In patients with Alzheimer's disease (AD) who respond to antipsychotic treatment of psychosis and/or agitation/aggression, the relapse risk after discontinuation is not established. AD patients with psychosis and/or agitation/aggression receive 16 weeks of open risperidone treatment (Phase A). Responders are then randomized, double-blind, to one of three arms in Phase B: (1) continuation risperidone for 32 weeks, (2) risperidone for 16 weeks followed by placebo for 16 weeks, (3) placebo for 32 weeks. The primary outcome is time to relapse of psychosis/agitation.

DETAILED DESCRIPTION:
This multicenter study (6 academic sites and 2 non-academic sites) involves treating AD patients (assisted living or nursing home patients, and outpatients) using an atypical antipsychotic, risperidone. In Phase A, 180 AD patients with psychosis and/or agitation/aggression receive open treatment with risperidone for 16 weeks. Responders are randomized, double-blind, to one of three arms in Phase B: (1) continuation risperidone for the next 32 weeks, (2) risperidone for the next 16 weeks followed by placebo for 16 weeks, or (3) placebo for the next 32 weeks. The primary hypothesis is that in the first 16 weeks of Phase B, relapse risk will be lower with continuation risperidone (Arms 1 + 2) compared to discontinuation on placebo (Arm 3). The secondary hypothesis is that in the second 16 weeks of Phase B, relapse risk will be lower with continuation risperidone (Arm 1) compared to discontinuation on placebo (Arm 2). For both randomized time periods, the proportions who relapse will be compared for interpretive support. This design provides useful data on the efficacy and side effects of longer term treatment with risperidone, and, in particular, critical information about the time to relapse and likelihood of relapse in patients switched from risperidone to placebo. This information is essential to guide the clinician toward optimal use of such medications in one of the most challenging types of patients: the AD patient with psychosis and/or agitation/aggression. The results of this study will also help to address Federal regulations urging early antipsychotic discontinuation in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Dementia, either sex, age 50-95 years
* Probable Alzheimer's disease
* Intellectual impairment present for at least 6 months
* Mini Mental State Exam (MMSE) score of 5-26 for outpatients and 2-26 for nursing home patients
* Availability of informant who has had direct contact with the patient for an average of at least once every week during the 3 months prior to study entry
* Meets Neuropsychiatric Inventory (NPI) criteria for either (1) psychosis, or (2) agitation/aggression
* Able to mobilize independently (if wheelchair-bound, the patient must be able to self-propel)
* Free of psychotropic medication (or able to tolerate washout) for at least 1 week prior to study entry. Low dose antidepressants and sedative/hypnotics allowed if they cannot be washed out and the dose remains stable for the study duration
* Expected to complete the study (including all efficacy evaluations) and be without major sensory impairment that would prevent participation in any aspect of the study

Exclusion Criteria:

* Current primary Axis I psychiatric disorder other than AD
* Substance abuse or dependence currently, or within the past year
* Dementia due to head trauma
* History of allergy to risperidone or intolerance to risperidone
* Diffuse Lewy body disease
* History of seizure disorder, infectious encephalitis, Parkinson's disease, central nervous system (CNS) neoplasm, tardive dyskinesia, stroke, transient ischemic attack (TIA) or uncontrolled atrial fibrillation
* Use of monoamine oxidase inhibitors (MAOIs) and unable to undergo 3-week washout; patients also may not take MAOIs for 2 weeks after completing the study
* In treatment with (a) depot antipsychotic within 2 weeks of the screening visit
* Untreated or incompletely treated hypothyroidism
* Active, unstable medical condition that requires active medication adjustment or surgery
* Need for electroconvulsive treatment (ECT)
* Significant risk for harm to themselves or others as a result of randomization to placebo
* History of malignant neoplasm during the last 5 years

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davangere P. Devanand, MD, Principal Investigator — NYSPI/Columbia University
Locations (7):
- United States (7):
  - Tuscaloosa VA Medical Center, Department of Psychiatry, Tuscaloosa, Alabama
  - WLA VA Medical Center/UCLA, Psychiatry, Los Angeles, California
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Mount Sinai School of Medicine, Alzheimer's Disease Research Center, New York, New York
  - New York State Psychiatric Institute, Columbia University, New York, New York
  - Medical University of South Carolina, North Charleston, South Carolina

REFERENCES:
- [Result] Devanand DP, Mintzer J, Schultz SK, Andrews HF, Sultzer DL, de la Pena D, Gupta S, Colon S, Schimming C, Pelton GH, Levin B. Relapse risk after discontinuation of risperidone in Alzheimer's disease. N Engl J Med. 2012 Oct 18;367(16):1497-507. doi: 10.1056/NEJMoa1114058. PMID 23075176
- [Derived] Patel AN, Lee S, Andrews HF, Pelton GH, Schultz SK, Sultzer DL, Mintzer J, de la Pena D, Gupta S, Colon S, Schimming C, Levin B, Devanand DP. Prediction of Relapse After Discontinuation of Antipsychotic Treatment in Alzheimer's Disease: The Role of Hallucinations. Am J Psychiatry. 2017 Apr 1;174(4):362-369. doi: 10.1176/appi.ajp.2016.16020226. Epub 2016 Nov 18. PMID 27855483
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/21407047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from memory clinics including Alzheimer Research Centers, geriatric psychiatry clinics, VA clinics, physician referrals and advertising.
Pre-assignment Details: 180 Patients with Alzheimer's disease (AD) & psychosis or agitation-aggression received open treatment with risperidone for 16 weeks in Phase A. Of 180 patients, 112 were responders and 110 were randomized in Phase B.
  Phase B: 110 responders were randomized, double-blind, to one of three arms in Phase B.
Groups:
- Arm 1: Risperidone-Risperidone: Phase A involved open flexible dose risperidone treatment for 16 weeks. At 16 weeks, non-responders exited the study. Responders were randomized, double-blind, to one of three arms in Phase B: (1) continuation risperidone for 32 weeks (Arm 1), (2) risperidone for 16 weeks followed by placebo for 16 weeks (Arm 2), (3) placebo for 32 weeks (Arm 3).
  Phase B Arm 1: Risperidone for 16 weeks followed by risperidone for 16 weeks; Risperidone open label flexible dose was administered at a dose of 0.25 to 3 mg daily for first 16 weeks; dose at 16 weeks then fixed for the randomized trial
- Phase B Arm 2: Risperidone-Placebo: Phase A involved open flexible dose risperidone treatment for 16 weeks. At 16 weeks, non-responders exited the study. Responders were randomized, double-blind, to one of three arms in Phase B: (1) continuation risperidone for 32 weeks (Arm 1), (2) risperidone for 16 weeks followed by placebo for 16 weeks (Arm 2), (3) placebo for 32 weeks (Arm 3).
  Phase B Arm 2: Risperidone for 16 weeks followed by placebo for 16 weeks;
- Phase B Arm 3: Placebo-Placebo: Phase A involved open flexible dose risperidone treatment for 16 weeks. At 16 weeks, non-responders exited the study. Responders were randomized, double-blind, to one of three arms in Phase B: (1) continuation risperidone for 32 weeks (Arm 1), (2) risperidone for 16 weeks followed by placebo for 16 weeks (Arm 2), (3) placebo for 32 weeks (Arm 3).
  Phase B Arm 3: Patients were randomized to placebo for 32 weeks.
Period: Phase B 1st 16 Weeks
Arm/Group | Arm 1: Risperidone-Risperidone | Phase B Arm 2: Risperidone-Placebo | Phase B Arm 3: Placebo-Placebo
Started | 32 (Risperidone 16 weeks.) | 38 (Risperidone 16 weeks.) | 40 (Placebo 16 weeks.)
Completed | 13 | 27 | 13
Not Completed | 19 | 11 | 27
Not completed — Lack of Efficacy | 14 | 8 | 24
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Moved, Unclear reasons | 2 | 3 | 2
Not completed — Death | 1 | 0 | 0
Period: Phase B 2nd 16 Weeks
Arm/Group | Arm 1: Risperidone-Risperidone | Phase B Arm 2: Risperidone-Placebo | Phase B Arm 3: Placebo-Placebo
Started | 13 (Risperidone for 16 weeks.) | 27 (Placebo for 16 weeks.) | 13 (Placebo for 16 weeks.)
Completed | 10 | 14 | 10
Not Completed | 3 | 13 | 3
Not completed — Lack of Efficacy | 1 | 12 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Moved; unclear reason | 1 | 0 | 0
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase B Arm 1: Risperidone-Risperidone; Phase B Arm 2: Risperidone -Placebo; Phase B Arm 3: Placebo-Placebo: Phase A involved open flexible dose risperidone treatment for 16 weeks. At 16 weeks, non-responders exited the study. Responders were randomized, double-blind, to one of three arms in Phase B: (1) continuation risperidone for 32 weeks (Arm 1), (2) risperidone for 16 weeks followed by placebo for 16 weeks (Arm 2), (3) placebo for 32 weeks (Arm 3). For patients receiving risperidone ≥ 2 mg daily at end-Phase A, assignment to placebo in Phase B required an initial one-week taper with sequential double-blind placebo substitution (e.g., one 2 mg tablet switched to one 1 mg tablet and then to one placebo tablet) to reduce antipsychotic physical withdrawal effects.
- Total: Total of all reporting groups
Arm/Group | Phase B Arm 1: Risperidone-Risperidone | Phase B Arm 2: Risperidone -Placebo | Phase B Arm 3: Placebo-Placebo | Total
Number analyzed (Participants) | 32 | 38 | 40 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 7
  >=65 years | 30 | 35 | 38 | 103
Age Continuous [Mean (Standard Deviation); unit: years] | 80.7 (7.9) | 79.1 (8.0) | 80.3 (7.7) | 80.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 24 | 66
  Male | 10 | 18 | 16 | 44
Region of Enrollment [Number; unit: participants]
  United States | 32 | 38 | 40 | 110

OUTCOME MEASURES:

1. Primary Outcome: Relapse by Study Week 32
Description: A relapse occurred in Phase B (post-randomization) if both of the following criteria were met:
  1. Increase in the Neuropsychiatric Inventory (NPI) core score of 30% or more OR a 5-point increase from the baseline NPI score at the end of Phase A
  2. A score of 6 (much worse) or 7 (very much worse) on the Clinical Global Impression-Change (CGI-C) at any visit.
Time Frame: 0-16 weeks in Phase B (16-32 weeks in study)
Population: Analysis was performed as per intention to treat (ITT) principles.
Measure: Number; unit: participants
Groups:
- Phase B Arm 1: Risperidone-Risperidone: 32 patients randomized to Phase B Arm 1 received continuation risperidone for another 32 weeks.
- Phase B Arm 2: Risperidone -Placebo: 38 patients randomized to Phase B Arm 2 received risperidone therapy for 16 weeks followed by placebo for 16 weeks.
  In Phase B, relapse required ≥ 30% increase or 5-point increase in NPI core scores from end-Phase A and a score of 6 (much worse) or 7 (very much worse) on the CGI-C.
- Phase B Arm 3: Placebo-Placebo: 40 patients randomized to Phase B Arm 3 received placebo for 32 weeks. For patients receiving risperidone ≥ 2 mg daily at end-Phase A, assignment to placebo in Phase B required an initial one-week taper with sequential double-blind placebo substitution (e.g., one 2 mg tablet switched to one 1 mg tablet and then to one placebo tablet) to reduce antipsychotic physical withdrawal effects.
  In Phase B, relapse required ≥ 30% increase or 5-point increase in NPI core scores from end-Phase A and a score of 6 (much worse) or 7 (very much worse) on the CGI-C.
Arm/Group | Phase B Arm 1: Risperidone-Risperidone | Phase B Arm 2: Risperidone -Placebo | Phase B Arm 3: Placebo-Placebo
Number analyzed (Participants) | 32 | 38 | 40
participants | 15 | 8 | 24
Statistical Analysis 1: Comparison: Phase B Arm 1: Risperidone-Risperidone vs Phase B Arm 2: Risperidone -Placebo vs Phase B Arm 3: Placebo-Placebo; The primary hypothesis of a difference in survival functions between the initial Phase B placebo (Arm 3) and risperidone continuation (Arms 1+2) conditions was tested in the primary analysis using the stratified Cox analysis. For descriptive purposes, the overall rate of relapse was assessed as the number of follow-up or for secondary interpretative support, as a simple proportion of patients entering a 16-week period; Test type: Superiority or Other; p = 0.02, Stratified Cox analysis; Hazard Ratio (HR) = 1.94, 95% CI 2-sided [1.09 to 3.45]

2. Secondary Outcome: Relapse by Study Week 48
Description: Same definition and criteria as the primary outcome
Time Frame: 16-32 weeks in Phase B (32-48 weeks in study)
Population: Randomized subjects in each Arm who had not relapsed or terminated the study by the end of the first 16 weeks of Phase B were analyzed in the second 16 weeks of Phase B using intent to treat (ITT) principles.
Measure: Number; unit: participants
Groups:
- Arm 1: Risperidone - Risperidone: Subjects in Arm 1 who did not relapse or terminate from the study in the first 16 weeks of Phase B continued to receive risperidone in the second 16 weeks of Phase B.
- Arm 2: Risperidone - Placebo: Subjects in Arm 2 who did not relapse or terminate from the study in the first 16 weeks of Phase B received placebo in the second 16 weeks of Phase B.
Arm/Group | Arm 1: Risperidone - Risperidone | Arm 2: Risperidone - Placebo
Number analyzed (Participants) | 13 | 27
participants | 2 | 13
Statistical Analysis 1: Comparison: Arm 1: Risperidone - Risperidone vs Arm 2: Risperidone - Placebo; Similar analyses were used to test the secondary hypothesis in the relapse risk in weeks 17 to 32 of Phase B between the patients who continued to receive risperidone (Arm 1) & the patients who discontinued risperidone at week 16 & were switched to placebo (Arm 2). Patients who died & those in whom a relapse was considered to be imminent before they were dropped out in Phase B were classified as having relapse; Test type: Superiority or Other; p = 0.02, stratified cox analyses; Hazard Ratio (HR) = 4.88, 95% CI 2-sided [1.08 to 21.98]

3. Secondary Outcome: Mini Mental State Exam (MMSE)
Description: The MMSE assesses cognition. Scores range from 0-30, with higher scores indicating better cognition. For each subject, the change in MMSE between week 16 and baseline (randomization) was calculated by subtraction, so that a positive value indicates an increase in MMSE over time.
Time Frame: Phase B, weeks 1-16 (study weeks 16-32)
Population: MMSE data were missing for 2 subjects in the placebo group and 1 subject in the risperidone group, so the number of subjects in this analysis were 38 (placebo) and 69 (risperidone), for a total of 107.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Subjects assigned to Arm 3, as described above
- Risperidone: Subjects in Arm 1 and Arm 2, as described above. Subjects in these two arms received risperidone for the first 16 weeks of Phase B, and were combined for purposes of this secondary analysis.
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 38 | 69
units on a scale | -0.13 (1.49) | -0.77 (2.23)
Statistical Analysis 1: Comparison: Placebo vs Risperidone; The null hypothesis is that there is no difference between the risperidone and placebo groups over the 16 week period post randomization, with respect to change in MMSE; Test type: Superiority or Other; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.08 to 1.35], Standard Error of Mean 0.36

4. Secondary Outcome: Treatment Emergent Symptoms Scale (TESS)
Description: The Treatment Emergent Symptom Scale (TESS) assesses 26 somatic symptoms. Total scores range from 0-26, with a score of 0 or 1 for each item. Higher scores indicate more somatic symptoms. For each subject, the change in TESS between week 16 and baseline (randomization) was calculated by subtraction, so that a positive value indicates an increase in TESS over time.
Time Frame: Phase B, weeks 1-16 (study weeks 16-32)
Population: All randomized subjects were included in this analysis (N=110)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 40 | 70
units on a scale | 0.18 (2.4) | 0.21 (2.5)
Statistical Analysis 1: Comparison: Placebo; The null hypothesis is that there is no difference between the risperidone and placebo groups over the 16 week period post randomization, with respect to change in TESS; Test type: Superiority or Other; p = 0.94, t-test, 2 sided; Mean Difference (Final Values) = -0.04, 95% CI [-1.01 to 0.93], Standard Error of Mean 0.49

5. Secondary Outcome: Extrapyramidal Signs (EPS)
Description: Extrapyramidal signs, also known as Parkinsonian signs, refer to signs of tremor, rigidity, and bradykinesia (slowed movement) that are seen in Parkinson's disease. Assessment of extrapyramidal signs (EPS) were made with the use of the Simpson-Angus scale (which ranges from 1-40) with higher scores indicating more extrapyramidal signs. For each subject, the change in EPS between week 16 and baseline (randomization) was calculated by subtraction, so that a positive value indicates an increase in EPS over time.
Time Frame: Phase B, weeks 1-16 (study weeks 16-32)
Population: All randomized subjects were included in the analysis (N=110).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 40 | 70
units on a scale | -0.20 (1.91) | 0.34 (2.68)
Statistical Analysis 1: Comparison: Placebo vs Risperidone; The null hypothesis is that the difference between placebo and risperidone groups in terms of mean change in EPS, between randomization and week 16, is zero; Test type: Superiority or Other; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.50 to 0.41], Standard Error of Mean 0.48

6. Secondary Outcome: AIMS
Description: The Abnormal Involuntary Movement Scale (AIMS) assesses signs of tardive dyskinesia, a movement disorder that can occur with prolonged use of antipsychotic medication. The AIMS score ranges from 0 to 35, with higher scores indicating more severe symptoms. For each subject, the change in AIMS score between week 16 and randomization was calculated by subtraction, so that a positive value indicates an increase in AIMS over time.
Time Frame: Phase B, weeks 1-16 (study weeks 16-32)
Population: All randomized subjects were included in this analysis (N=110).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 40 | 70
units on a scale | 0.03 (0.48) | 0.24 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Risperidone; The null hypothesis is that the difference between placebo and risperidone groups in terms of mean change in AIMS, between randomization and week 16, is zero; Test type: Superiority or Other; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.50 to 0.07], Standard Error of Mean 0.14

7. Secondary Outcome: Physical Self-Maintenance Scale (PSMS)
Description: Physical Self-Maintenance Scale, which ranges from 1 to 30, with higher scores indicating WORSE functioning. For each subject, the change in PSMS between week 16 and randomization was calculated by subtraction, so that a positive value indicates an increase in PSMS (worse functioning) over time.
Time Frame: Phase B, weeks 1-16 (study weeks 16-32)
Population: All randomized subjects were included in this analysis, with the exception of one placebo subject for whom PSMS data was not available at one time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 39 | 70
units on a scale | 0.18 (1.73) | 0.80 (2.72)
Statistical Analysis 1: Comparison: Placebo vs Risperidone; The null hypothesis is that the difference between placebo and risperidone groups in terms of mean change in PSMS, between randomization and week 16, is zero; Test type: Superiority or Other; p = 0.149, t-test, 2 sided; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.47 to 0.23], Standard Error of Mean 0.43

8. Secondary Outcome: Weight
Description: For each subject, the change in weight in pounds between week 16 and randomization was calculated by subtraction, so that a positive value indicates an increase in weight over time.
Time Frame: Phase B, weeks 1-16 (study weeks 16-32)
Population: Available data from all randomized subject (N=110) was used in this analysis. Weight measurements were unavailable at one or more time points for 3 subjects in the placebo group and for 6 subjects in the risperidone group.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 37 | 64
pounds | 0.32 (7.18) | 0.73 (8.71)
Statistical Analysis 1: Comparison: Placebo vs Risperidone; The null hypothesis is that the difference between placebo and risperidone groups in terms of mean change in weight, between randomization and week 16, is zero; Test type: Superiority or Other; p = 0.81, t-test, 2 sided; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-3.77 to 2.95], Standard Error of Mean 1.69

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial, in both the open treatment Phase A (study week 1-16) and in the post-randomization Phase B (study weeks 16-48)
Groups:
- Wk0-16 Phase B Arm 1 (Risp-Risp) & Arm 2 (Risp-Pla): 32 patients randomized to Phase B Arm 1 received continuation risperidone for another 32 weeks; 38 patients randomized to Phase B Arm 2 received risperidone for 16 weeks followed by placebo for 16 weeks. Therefore there were a total of 70 patients in this group.
- Wk 0-16 Phase B Arm 3: Placebo -Placebo: 40 patients randomized to Phase B Arm 3 received placebo for 32 weeks.
- Wk 17-32 Phase B Arm 1: Risperdone-Risperdone: 13 patients completed Wk 0-16 of Phase 2 Arm 1 and entered Wk 17-32 where they received risperidone for another 16 weeks.
- Wk 17-32 Phase B Arm 2: Risperdone-Placebo: 27 patients completed Wk 0-16 of Phase B Arm 2 and entered Week 17-32 of Phase B Arm 2 where they receive placebo for 16 weeks.
- Wek 17-32 Phase B Arm 3: Placebo -Placebo: 13 patients completed Week 0-16 of Phase B Arm 3 and entered Week 17-32 were they were given placebo for another 16 weeks.
Arm/Group | Wk0-16 Phase B Arm 1 (Risp-Risp) & Arm 2 (Risp-Pla) | Wk 0-16 Phase B Arm 3: Placebo -Placebo | Wk 17-32 Phase B Arm 1: Risperdone-Risperdone | Wk 17-32 Phase B Arm 2: Risperdone-Placebo | Wek 17-32 Phase B Arm 3: Placebo -Placebo
Serious Adverse Events (participants affected / at risk) | 5/70 | 8/40 | 2/13 | 0/27 | 0/13
Other Adverse Events (participants affected / at risk) | 36/70 | 24/40 | 9/13 | 13/27 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wk0-16 Phase B Arm 1 (Risp-Risp) & Arm 2 (Risp-Pla) (N=70) | Wk 0-16 Phase B Arm 3: Placebo -Placebo (N=40) | Wk 17-32 Phase B Arm 1: Risperdone-Risperdone (N=13) | Wk 17-32 Phase B Arm 2: Risperdone-Placebo (N=27) | Wek 17-32 Phase B Arm 3: Placebo -Placebo (N=13)
Death (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular Event (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neurologic Event (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation-Aggression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall or Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wk0-16 Phase B Arm 1 (Risp-Risp) & Arm 2 (Risp-Pla) (N=70) | Wk 0-16 Phase B Arm 3: Placebo -Placebo (N=40) | Wk 17-32 Phase B Arm 1: Risperdone-Risperdone (N=13) | Wk 17-32 Phase B Arm 2: Risperdone-Placebo (N=27) | Wek 17-32 Phase B Arm 3: Placebo -Placebo (N=13)
Extrapyramidal signs (Nervous system disorders) | 13 (13) | 4 (4) | 4 (4) | 4 (4) | 2 (2) — Extrapyramidal signs was considered to be adverse events if there was an average increase from baseline of more than 1 point on the Simpson-Angus scale.
akathisia or restlessness (Nervous system disorders) | 4 (4) | 6 (6) | 1 (1) | 3 (3) | 1 (1) — Akathisia or restlessness was considered to be adverse events if there was an average increase from baseline of more than 1 point on the Simpson-Angus scale.
sedation (Nervous system disorders) | 7 (7) | 5 (5) | 1 (1) | 1 (1) | 1 (1) — Sedation was either a report of clinically significant new adverse event or a worsening of a symptom from baseline to a moderate or severe level, as assessed by means of the Treatment Emergent Symptom scale (TESS).
insomnia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Insomnia was either a report of clinically significant new adverse event or a worsening of a symptom from baseline to a moderate or severe level, as assessed by means of the Treatment Emergent Symptom scale (TESS).
confusion (Nervous system disorders) | 4 (4) | 4 (4) | 1 (1) | 3 (3) | 1 (1) — Confusion was either a report of clinically significant new adverse event or a worsening of a symptom from baseline to a moderate or severe level, as assessed by means of the Treatment Emergent Symptom scale (TESS).
Agitation-Aggression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Agitation-aggression was either a report of clinically significant new adverse event or a worsening of a symptom from baseline to a moderate or severe level, as assessed by means of the Treatment Emergent Symptom scale (TESS).
fall (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Fall was either a report of clinically significant new adverse event or a worsening of a symptom from baseline to a moderate or severe level, as assessed by means of the Treatment Emergent Symptom scale (TESS).
nausea or vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) — Nausea or vomiting was either a report of clinically significant new adverse event or a worsening of a symptom from baseline to a moderate or severe level, as assessed by means of the Treatment Emergent Symptom scale (TESS).

LIMITATIONS AND CAVEATS:
Comparisons of adverse events in Phase B were limited by the small sample & the truncated observation period for relapsed subjects. Identification of predictors of relapse after discontinuation of treatment was limited by the small sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No